CLINICAL TRIAL: NCT03299127
Title: A Self-help Manual of Imagery Rescripting Reduces Depressive Symptoms
Brief Title: Imagery Rescripting in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR-Phoenix
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: randomized-controlled trial, wait-list control condition
Masking Description: self-report serves as outcomes, patients are not masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- imagery rescripting (Experimental): bibliotherapy, intervention is provided by pdf-manual (either short or long version, i.e. 2 active arms, each 1/3 of sample receives either short or long version)
  Interventions: Behavioral: imagery rescripting
- wait-list control (No Intervention): wait-list control, participants receive intervention manual upon completion of post-assessment (1/3 of sample)

INTERVENTIONS:
Behavioral: imagery rescripting — The long version of the manual contained 4,959 words, the brief version had 3,369 words. Individuals were encouraged patients to time travel to negative personal events, enter the scene and protect or comfort their younger-ego. The participant should bring the negative event to a "happy end. This could also be a fictive, compassionate person and may violate the laws of physics (e.g., a person may fly). Readers were encouraged to embellish the scenes as much as possible so that it competed with the original scene. This technique was then applied to future events. For the last technique, patients were asked to seek a corresponding mood-congruent metaphor, creature or symbol; for example, a small bird that has fallen out of its nest. Using their mind's eye, these images may be transformed into something of beauty or pride.
  Arms: imagery rescripting

SUMMARY:
Depression is among the world's leading causes of disability. To fill the existing treatment gap, psychological online interventions (POIs) and Internet-based treatment, including bibliotherapy with PDF manuals (POIs), are increasingly recommended as they are easily accessible and deemed an initial alternative approach. The present trial aims to evaluate imagery rescripting. With the help of various techniques, the approach aims to edit negative memories and rewrite a "happy end". To the best of our knowledge, imagery rescripting has never been tested as a self-help intervention. A large sample of patients with primary or secondary depression (N = 120) will be recruited and randomly allocated to either the intervention group or a wait-list control group. The intervention group consists of two subgroups that will receive either a full or brief version of a manual teaching them imagery rescripting. Participants will be assessed at baseline and six weeks later. A follow-up assessment will be completed six months later. The primary outcome measure is the Beck Depression Inventory II.

DETAILED DESCRIPTION:
Depression is among the world's leading causes of disability. Effective pharmacological and psychotherapeutic treatments exist. However, only a subgroup of individuals with depressive symptoms receive proper treatment (Kohn, Saxena, Levav, & Saraceno, 2004). To fill the existing treatment gap (Kazdin, 2017), psychological online interventions (POIs) and Internet-based treatment, including bibliotherapy with PDF manuals (POIs), are increasingly recommended as they are easily accessible and deemed an initial alternative approach (i.e., "foot in the door") for persons who have reservations about face-to-face psychotherapy. E-mental health and bilbiotherapeutic interventions have yielded promising results, but there remains room for improvement as effect sizes are usually in the small to medium range. The present trial aims to evaluate imagery rescripting, a technique developed by Smucker (Smucker, Dancu, Foa, & Niederee, 1995). With the help of various techniques, the approach aims to edit negative memories and rewrite a "happy end". Positive mental imagery strategies seek to hold negative mental images in check and impart the patient with a feeling of self-efficacy. A new meta-analysis shows that imagery rescripting yields large effects on anxiety and depressive symptoms across a range of disorders (Morina, Lancee, & Arntz, 2017).

To the best of our knowledge, imagery rescripting has never been tested as a self-help intervention. A large sample of patients with primary or secondary depression (N = 120) will be recruited and randomly allocated to either the intervention group or a wait-list control group. The intervention group consists of two subgroups that will receive either a full or brief version of a manual teaching them imagery rescripting. Participants will be assessed at baseline and six weeks later. At post-assessment, the (full-length) manual will be made available to all participants. A follow-up assessment will be completed six months later. The primary outcome measure is the Beck Depression Inventory II. Secondary outcome measures include self-reported symptom measures (PHQ-9, GAF-7, Rosenberg Self-Esteem Scale, Global item from the WHOQOL-BREF). The project may help to answer the question of whether imagery rescripting is effective when presented using a self-help medium.

ELIGIBILITY:
Inclusion Criteria:

* Electronic informed consent
* Internet access
* Adequate command of the German language
* Diagnosis of depression (primary or secondary)

Exclusion Criteria:

* Acute suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory II | Change in BDI-II from pre- to post-intervention (i.e. 6 week interval)
  Beck Depression Inventory II (BDI II) (Beck, Steer, & Brown, 1996). The BDI-II is a self-report scale that contains 21 Items that tap into cognitive, behavioral and somatic symptoms of depression. A follow-up assessment after six month serves as secondary outcome.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Change from pre- to post-intervention (i.e. 6 week interval)
  The Patient Health Questionnaire (PHQ-9) is a self-administered scale derived from the Primary Care Evaluation of Mental Disorders (PRIME-MD) and measures depression according to the nine depression items of the DSM-IV.
Rosenberg Self-Esteem Scale (RSE) | Change from pre- to post-intervention (i.e. 6 week interval)
  The Rosenberg Self-Esteem Scale (RSE) assesses self-esteem with 10 items.
Generalized Anxiety Disorders 7 (GAD-7) | Change from pre- to post-intervention (i.e. 6 week interval)
  The Generalized Anxiety Disorders 7 (GAD-7) is a screening instrument for common anxiety symptoms consisting of seven items.
Global item of the WHO Quality of Life scale (WHOQOL-BREF) | Change from pre- to post-intervention (i.e. 6 week interval)
  The global item of the WHO Quality of Life scale (WHOQOL-BREF) assesses quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Moritz, PhD, Principal Investigator — UKE Hamburg
Locations (1):
- University Medical Center Hamburg Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Moritz S, Ahlf-Schumacher J, Hottenrott B, Peter U, Franck S, Schnell T, Peter H, Schneider BC, Jelinek L. We cannot change the past, but we can change its meaning. A randomized controlled trial on the effects of self-help imagery rescripting on depression. Behav Res Ther. 2018 May;104:74-83. doi: 10.1016/j.brat.2018.02.007. Epub 2018 Feb 26. PMID 29597112